CLINICAL TRIAL: NCT02900352
Title: Zonisamide Treatment of Alcohol Use Disorder: an Evaluation of Efficacy and Mechanism of Action
Acronym: Z-Comp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Connecticut (Other); Yale University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20014185; 1605017700 (Other: Yale University); 7R01AA024466-04 (NIH)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Alcoholism; Alcohol Dependence; Zonisamide; Alcohol Intoxication; Drinking Behaviors; Anticonvulsants
MeSH Terms: conditions — Alcoholism; Alcoholic Intoxication; Drinking Behavior | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zonisamide (Experimental): Subjects will receive zonisamide titrated to a target dose of 500mg orally, daily, double-blind (Titration of dose to 500mg oral, daily, over 7 weeks, then 9 weeks of treatment at that dose). Subjects may increase their dose to 600mg daily during the target treatment period if it is thought to be beneficial.
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator): Patients will receive placebo pills that are made to match the zonisamide medication (via over-encapsulation, double-blind, subjects will receive same number of capsules as the active medication group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose
  Other Names: Brand name: Zonegran
  Arms: Zonisamide
Drug: Placebo — Placebo
  Other Names: Brand name: Zonegran
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 16 week trial of the medication zonisamide for the treatment of heavy drinking alcoholic civilians.

DETAILED DESCRIPTION:
This is a 16-week randomized, double blind, placebo-controlled trial designed to determine the effectiveness of zonisamide treatment for reducing heavy drinking and overall drinking in 160 treatment-seeking, regularly heavy drinking, alcohol-dependent civilians who want to quit drinking or reduce consumption to non-hazardous levels. The investigators will use state-of-the-art methodology and outcome assessments, including medical management (MM) therapy (a minimal behavioral intervention aimed at reinforcing treatment goals and adherence to medication), which is simple and easily implemented in primary care settings. The use of MM in the study will increase the generalizability of results, allowing a more accurate assessment of zonisamide's effectiveness than if a more intensive behavioral intervention were to be used. To demonstrate zonisamide's effectiveness in a representative civilian sample, the investigators will include civilians with co-morbid mood and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Female/male aged 21-70 years
* Regular heavy drinkers as defined by averaging 2 heavy drinking days per week over 90 days baseline pre-treatment timeline follow-back (TLFB), and current DSM-IV-TR alcohol dependence that recognize a need to reduce or stop drinking (Note: heavy drinking days will be defined as follows; for men greater than or equal to 5 drinks in a day and for women greater than or equal to 4 drinks in a day)
* Women of child-bearing potential (i.e., no hysterectomy, bilateral oophorectomy, or tubal ligation or <2 years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment;
* Willingness to provide signed, informed consent to participate in the study

Exclusion Criteria:

* A current, clinically significant physical disease or abnormality (i.e., neurologic, renal, rheumatologic, gastrointestinal, hematologic, pulmonary, endocrine, cardiovascular, hepatic, or autoimmune disease that, in the context of the study would represent a risk to the subject, or significant laboratory abnormalities such as hepatic aminotransferase levels (i.e., AST and ALT) greater than 300% of the upper limit of normal or direct bilirubin levels >150% of the upper limit of normal) on the basis of medical history, physical examination, or routine laboratory evaluation. Other specific exclusionary disorders include;
* History of clinically significant renal calculi or renal failure; a significant indication of renal compromise will be defined by an elevation of serum creatinine above the investigators' laboratory's limit of normal, or a known history of renal failure or chronic renal disease, or any current or chronic disease that could reasonably be expected to result in renal failure
* History of hypersensitivity to ZNS or any sulfonamide, Stevens-Johnson Syndrome, penicillin allergy, or history of any severe drug allergic reaction; History of systemic autoimmune disease such as lupus erythematosis, fibromyalgia, or rheumatoid arthritis;
* Current blood dyscrasia or a history of such, with the exception of a past history of iron deficiency anemia
* History of seizure disorder
* Use of any of a number of medications that might prominently influence drinking patterns or cause risk of harm or injury (e.g., topiramate, disulfiram, naltrexone, acetazolamide, stimulants such as amphetamine, or tramadol; Schizophrenia, bipolar disorder, PTSD, or substantial suicide or violence risk (i.e., can't be managed safely in the outpatient setting) on the basis of history or psychiatric examination; j) currently dependent on opioids or benzodiazepines or other sedatives
* Considered by the investigators to be clinically inappropriate for study participation or have participated in another pharmacotherapy study in the past thirty days
* Subjects with prominent signs of physical dependence, and/or medical comorbidities such that study physicians feel they should consider immediate detoxification, and referred for medical detoxification in a normal treatment setting

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-10; Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Arias, MD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - UCONN Health, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - West Haven Veterans Affairs, West Haven, Connecticut
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 77 | 79
Completed | 49 | 62
Not Completed | 28 | 17
Not completed — Lost to Follow-up | 28 | 17

BASELINE CHARACTERISTICS:
Population: Alcohol Use Disorder Treatment Seekers
Groups:
- Zonisamide: Subjects will receive zonisamide titrated to a target dose of 500mg orally, daily, double-blind (Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose). Subjects may increase their dose to 600mg daily during the target treatment period if it is thought to be beneficial.
  Zonisamide: Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 77 | 79 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.6) | 51.9 (9.7) | 51.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 46 | 52 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 70 | 75 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 63 | 66 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 77 | 79 | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Per Week
Description: Difference between groups in the number of total standard drinks per week over 8 weeks (weeks 9-16, the weeks on the target dose) performed using a mixed models longitudinal analysis.
Time Frame: over 8 weeks (weeks 9-16)
Measure: Mean (Standard Error); unit: Number of drinks per week
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 77 | 79
Number of drinks per week | 19.7 (2.2) | 23.7 (1.98)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.0130, Mixed Models Analysis

2. Secondary Outcome: Percentage of Subjects With No Heavy Drinking Days
Description: percentage of subjects with no heavy drinking days (PSNHDD) The PSNHDD can be derived from each subject's Timeline Followback (TLFB) data.
Time Frame: over the last 8 weeks (weeks 9-16)
Measure: Number; unit: Percentage of participants
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 77 | 79
Percentage of participants | 8.97 | 5.13
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.148, Chi-squared

3. Secondary Outcome: Gamma Glutamyl Transferase (GGT) Levels
Description: Difference between groups on levels of GGT over time from baseline to endpoint, which will includes two interim data points for a total of four time points. This will analyzed with a mixed models longitudinal analysis (repeated measures). Levels are in Units per Liter.
Time Frame: over 16 weeks (weeks 1-16)
Population: Due to protocol changes over the course of the study, data for some outcomes was not collected for all participants or collected at slightly different timepoints. Results are reported for all participants for whom data is available.
Measure: Mean (Standard Error); unit: International Units per Liter (UI/L)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 74 | 77
International Units per Liter (UI/L)
  Baseline Visit | 78.35 (12.10) | 71.88 (11.12)
  Visit 5 (Week 5): number analyzed (Participants) | 12 | 15
  Visit 5 (Week 5) | 52.33 (23.7) | 64.4 (29.35)
  Visit 7 (Week 9): number analyzed (Participants) | 53 | 58
  Visit 7 (Week 9) | 59.49 (10.05) | 70.24 (24.43)
  Visit 9 (Week 13): number analyzed (Participants) | 1 | 4
  Visit 9 (Week 13) | 16.0 (0.0) | 25.75 (5.75)
  Visit 10 (Week 16): number analyzed (Participants) | 42 | 51
  Visit 10 (Week 16) | 54.48 (7.83) | 56.65 (10.23)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = .054, ANOVA

4. Secondary Outcome: Number of Heavy Drinking Days Per Week
Description: The difference in the number of heavy drinking days per week compared between groups (zonisamide and placebo) for the last 8 weeks of treatment (during the time spent on the target dose of the medication). Performed using a mixed models longitudinal analysis (repeated measures).
Time Frame: over the last 8 weeks (weeks 9-16)
Population: Due to protocol changes over the course of the study, data for some outcomes was not collected for all participants. Results are reported for all participants for whom data is available.
Measure: Mean (Standard Error); unit: Number of heavy drinking days/week
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 59 | 71
Number of heavy drinking days/week | 2.7 (.34) | 3.3 (.30)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.035, Mixed Models Analysis

5. Secondary Outcome: Change in Alcohol Urge Questionnaire Score (AUQ)
Description: This is the change in AUQ scores (urge to drink) measured weekly compared between groups using repeated measures
  Min value: 8 Max value: 42 higher score = worse craving
Time Frame: over 16 weeks (weeks 1-16) and at 2 week and 3 month follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 58 | 67
score on a scale
  Visit 2 (Baseline) | 16.2 (1.04) | 16.06 (1.04)
  Visit 3 (Week 1) | 14.4 (0.96) | 17.12 (1.2)
  Visit 4 (Week 3) | 15.2 (1.12) | 15.28 (0.96)
  Visit 5 (Week 5) | 13.84 (1.09) | 14.4 (1)
  Visit 6 (Week 7) | 12.8 (0.96) | 14.72 (1.04)
  Visit 7 (Week 9) | 14.08 (1.2) | 16.24 (1.12)
  Visit 8 (Week 11) | 13.6 (1.2) | 14.56 (1.12)
  Visit 9 (Week 13) | 13.6 (1.2) | 14.4 (0.96)
  Visit 10 (Week 16) | 13.36 (1.2) | 13.36 (.96)
  Visit 11 (2 Week follow up) | 14.56 (.17) | 14.32 (1.04)
  Visit 12 (3 Month follow up) | 14.16 (1.28) | 13.68 (.96)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.889, ANOVA

6. Secondary Outcome: Change in Quality of Life
Description: Change in quality of life scores measured by the Q-LES-Q. ' Min: 16 Max: 80 Higher Scores = Higher Life Enjoyment
Time Frame: over 16 weeks (weeks 1-16) and at 2 week and 3 month follow up
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 60 | 60
score on a scale
  Visit 2 (Baseline) | 60 (13.6) | 59.84 (12.48)
  Visit 10 (Week 16): number analyzed (Participants) | 46 | 51
  Visit 10 (Week 16) | 61.6 (1.6) | 63.2 (13.44)
  Visit 11 (2 Week Follow up) | 68 (2.96) | 60.48 (2.72)
  Visit 12 (3 Month Follow up): number analyzed (Participants) | 35 | 46
  Visit 12 (3 Month Follow up) | 65.12 (12.96) | 64.64 (13.76)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.482, ANOVA

7. Secondary Outcome: Level of Alcohol-related Problems
Description: level of alcohol-related problems measured by the Short Index of Problems (SIP), total score
  Min score: 0 Max Score: 45 Higher score= more problems
Time Frame: over 16 weeks (weeks 1-16) and at 2 week and 3 month follow up
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 50 | 58
score on a scale
  Visit 2 (Baseline) | 14.94 (1.13) | 16.4 (.94)
  Visit 10 (Week 16) | 8.32 (1.23) | 11.6 (1.03)
  Visit 12 (3 Month follow up) | 6.92 (1.08) | 9.69 (1.18)
Statistical Analysis 1: Comparison: Zonisamide vs Placebo; Test type: Superiority; p = 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: Duration of the study (16 weeks)
Description: Patients provided subjective reports of side effects at each study visit using the Systematic Assessment for Treatment Emergent Effects (SAFTEE) interview, a widely used measure of adverse events. Complex adverse events may have also been recorded using non-systematic methods
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 1/79
Serious Adverse Events (participants affected / at risk) | 2/77 | 2/79
Other Adverse Events (participants affected / at risk) | 73/77 | 76/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=77) | Placebo (N=79)
Stroke (Cardiac disorders) | 1 (1) | 0 (0) — 1 participant (ppt) experienced stroke during study. Medication was tapered, blind was broken, ppt was withdrawn from study.
Alcohol Withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — 1 ppt had voluntarily requested treatment for detoxification. Ppt was admitted to 5 day inpatient alcohol detox.
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — 1 ppt died in MVA while travelling out of state. Not study related and was on placebo. This incident was reported to the UConn IRB and Dr. Arias
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — 1 ppt contacted study team to report suicidal ideation and possible attempt, they were assessed at a hospital and discharged home, were tapered off study medication and follow-up engaged in outpatient clinic.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=77) | Placebo (N=79)
Abdominal Pain (Gastrointestinal disorders) | 15 (22) | 13 (24)
Nausea (Gastrointestinal disorders) | 17 (30) | 11 (19)
Vomiting (Gastrointestinal disorders) | 9 (11) | 6 (7)
Extreme Tiredness (Nervous system disorders) | 24 (62) | 22 (44)
Constipation (Gastrointestinal disorders) | 9 (30) | 11 (20)
Diarrhea (Gastrointestinal disorders) | 11 (44) | 8 (53)
Nervousness (Psychiatric disorders) | 6 (10) | 13 (28)
Feeling Drowsy (Psychiatric disorders) | 22 (53) | 15 (42)
Fatigue (Psychiatric disorders) | 28 (81) | 23 (69)
Depressed Mood (Psychiatric disorders) | 22 (61) | 22 (58)
Swelling or Puffiness (Skin and subcutaneous tissue disorders) | 5 (11) | 7 (14)
Nasal Congestion/Runny Nose (Respiratory, thoracic and mediastinal disorders) | 36 (96) | 36 (128)
Rash or Skin Problem (Skin and subcutaneous tissue disorders) | 14 (29) | 13 (35)
Ringing in Ears (Nervous system disorders) | 8 (16) | 15 (60)
Decreased Sex Drive (Reproductive system and breast disorders) | 7 (22) | 13 (42)
Impotence (Reproductive system and breast disorders) | 4 (12) | 7 (27)
Headache (Nervous system disorders) | 17 (32) | 21 (48)
Blurred Vision (Eye disorders) | 6 (8) | 7 (25)
Gas (Gastrointestinal disorders) | 7 (7) | 6 (6)
Feeling dizzy, faint, lightheaded (Nervous system disorders) | 1 (1) | 4 (4)
Back, Muscle, or Bone Pain (Musculoskeletal and connective tissue disorders) | 26 (87) | 34 (103)
Mood Swings (Psychiatric disorders) | 8 (10) | 9 (28)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 7 (28)
Loss of Appetite (Gastrointestinal disorders) | 16 (38) | 9 (31)
Difficulty Sleeping (Psychiatric disorders) | 33 (107) | 36 (132)
Teary or Dry Eyes (Eye disorders) | 10 (24) | 13 (34)
Extreme Thirst (Gastrointestinal disorders) | 8 (11) | 8 (13)
Heartburn (Gastrointestinal disorders) | 16 (49) | 15 (51)
Memory Problems (Psychiatric disorders) | 12 (26) | 9 (20)
Difficulty concentrating or paying attention (Pregnancy, puerperium and perinatal conditions) | 17 (32) | 13 (45)
Numbness or Tingling around Mouth, Fingers, or Toes (Nervous system disorders) | 20 (48) | 15 (45)
Swelling of Feet or Ankles (Skin and subcutaneous tissue disorders) | 5 (13) | 8 (22)
Restlessness, Can't sit still (Psychiatric disorders) | 11 (16) | 12 (18)
Anger or Irritability (Psychiatric disorders) | 11 (27) | 21 (43)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 8 (9) | 15 (37)
Itching (Skin and subcutaneous tissue disorders) | 13 (30) | 10 (38)
Dry Mouth (Gastrointestinal disorders) | 14 (32) | 10 (26)
Unusual Sensations on Skin (Nervous system disorders) | 5 (8) | 8 (21)
Fever (General disorders) | 5 (10) | 3 (3)
Chills (General disorders) | 7 (9) | 4 (6)
Problems with Urination (Renal and urinary disorders) | 6 (6) | 5 (5)
Gas (Gastrointestinal disorders) | 17 (37) | 13 (45)
Irregular Heartbeat (Cardiac disorders) | 4 (4) | 2 (3)
Feeling Dizzy, Faint, or Lightheaded (General disorders) | 11 (16) | 15 (26)
Weakness (General disorders) | 4 (7) | 4 (18)
Trouble Walking (General disorders) | 6 (8) | 10 (29)
Hair Loss (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Confusion or Slowed Thinking (Psychiatric disorders) | 9 (17) | 10 (22)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (14)
Trouble Breathing (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 4 (15)
Change in Ability to Taste Food (Gastrointestinal disorders) | 9 (10) | 3 (5)
Tremors or Shakiness (Nervous system disorders) | 4 (5) | 5 (5)
Trouble with Gums (General disorders) | 3 (8) | 4 (4)
Sore Throat (Gastrointestinal disorders) | 6 (9) | 11 (13)
Unusual Bruising or Bleeding (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
Double Vision or Changes In Vision (Eye disorders) | 1 (7) | 6 (8)
Weight Loss (General disorders) | 8 (20) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02900352/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT02900352/ICF_001.pdf